CLINICAL TRIAL: NCT06707792
Title: Investigation of Validity and Reliability of 6 Minute Stepper Test in Kidney Transplant Recipients
Brief Title: Validity and Reliability of 6 Minute Stepper Test in Kidney Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: GO 23/604
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplanted Recipients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney transplant recipients

SUMMARY:
The aim of our study was to investigate the validity and reliability of the 6 minute stepper test in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney transplantation
* At least 6 months after the kidney transplant
* Not having regular exercise habits
* Voluntary participation in the study

Exclusion Criteria:

* Having a musculoskeletal problem that may interfere with the tests
* Having neurological impairment
* Having chronic lung disease
* Having had any cardiovascular event in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Day 1
  Exercise capacity will be assessed with a 6 minute stepper test.
Exercise capacity | Day 1
  Exercise capacity will be assessed with a 6 minute walk test.
Peripheral muscle strength | Day 1
  Knee extensor strength will be measured using a portable portable handheld dynamometer.
Lower extremity endurance | Day 1
  It will be evaluated with a one-minute sit to stand test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)